CLINICAL TRIAL: NCT03251898
Title: Multicenter Study on Correlation Between Premature Rupture of Membranes and Early-onset Neonatal Infections
Brief Title: Correlation Between Premature Rupture of Membranes and Early-onset Neonatal Infections
Status: Completed | Type: Observational
Sponsor: Bayi Children's Hospital Affiliated to PLA Army General Hospital, China (Other)
Collaborators: Northwest Women's and Children's Hospital, Xi'an, Shaanxi (Other); Chengdu Women's and Children's Central Hospital (Other); Shenzhen Maternity & Child Healthcare Hospital (Other); Nanjing Maternity and Child Health Care Hospital (Other); Shenzhen Bao'an Maternal and Child Health Hospital (Other); Second Hospital of Jilin University (Other)
Responsible Party: Sponsor
Organization: Seventh Medical Center of PLA General Hospital (Other)
Other Study IDs: BayiChildrens-01
Record Dates: First submitted 2017-08-15; First posted 2017-08-16 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2017-08

CONDITIONS: Premature Rupture of Membrane; Neonatal Infection
MeSH Terms: conditions — Fetal Membranes, Premature Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: pregnant women who are diagnosed as PROM or chorioamnionitis and whose gestational age is ≥ 24 weeks
- control group: pregnant women without PROM and chorioamnionitis

SUMMARY:
This study hypothesizes that early-onset neonatal Infections are related to premature rupture of membrane (PROM) and that early intervention can improve the prognosis of newborns. The objective of this study is to analyze the correlation between PROM and early-onset neonatal infections and to assess the prognosis of newborns. A cohort study is designed to implement the study. The subjects of study group are pregnant women who are diagnosed as PROM or chorioamnionitis and whose gestational age is ≥ 24 weeks. The subjects of control group are pregnant women without PROM and chorioamnionitis. Control group and research group are paired at 1: 1 ratio. The main contents of the study include three aspects. (1) The correlation between PROM and chorioamnionitis. (2) The correlation between PROM and early-onset neonatal infections. (3) The pathogenesis of intrauterine infection and neonatal infection.

ELIGIBILITY:
Inclusion Criteria:

* PROM or chorioamnionitis
* gestational age is ≥ 24 weeks

Exclusion Criteria:

* gestational age <24 weeks
* artificial rupture of membrane for labor induction
* natural rupture of membrane during induction before labor

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The pregnant women who are hospitalized to delivery in the collaborator hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 15926 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
the incidence of early-onset neonatal infections | 7 days after birth
  The incidence of early-onset neonatal infections will be compared between study group and control group.

CONTACTS AND LOCATIONS:
Overall Officials: Xing Li, Principal Investigator — Bayi Children's Hospital Affiliated to PLA Army General Hospital, China; Shaodong Hua, Principal Investigator — Bayi Children's Hospital Affiliated to PLA Army General Hospital, China; Jie Cui, Principal Investigator — Bayi Children's Hospital Affiliated to PLA Army General Hospital, China; Lei Li, Principal Investigator — Bayi Children's Hospital Affiliated to PLA Army General Hospital, China
Locations (6):
- China (6):
  - Chengdu Women's and Children's Central Hospital, Chengdu
  - Second Hospital of Jilin University, Jilin
  - Nanjing Maternity and Child Health Care Hospital, Nanjing
  - Shenzhen Bao'an Maternal and Child Health Hospital, Shenzhen
  - Shenzhen Maternity & Child Healthcare Hospital, Shenzhen
  - Northwest Women's and Children's Hospital, Xi'an